CLINICAL TRIAL: NCT02185742
Title: Planning for Sustained, Unbroken Connections to Care, Entry Services, and Suppression (SUCCESS)-- A Project to Improve the Connection to Community Care for HIV Infected Persons Leaving Jail in Atlanta
Brief Title: Planning for SUCCESS
Acronym: SUCCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Anne C Spaulding, Assoc Professor, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00064852; 1R34DA035728-01A1 (NIH)
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: HIV
Keywords: HIV; jail; detainee; Linkage and Retention; Treatment as Prevention; Strength Based Case Management; releases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strength Based Case Management (Experimental): Strength Based Case Management
  Interventions: Behavioral: Strength Based Case Management
- Contemporary, HIV+ Jail Detainees (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Strength Based Case Management
  Arms: Strength Based Case Management

SUMMARY:
Planning for SUCCESS (Sustained, Unbroken Connections to Care, Entry Services, and Suppression) is a project to improve the connection to community care for HIV infected persons leaving Fulton County Jail or Atlanta City Detention Center in Atlanta.

Hypothesis: Participants who receive the intervention will be more likely to link to medical care after jail release than similar participants who do not receive the intervention.

Rationale and objective: This project aims to make sure HIV positive persons leaving jail maintain medical care. Case managers will use strength based case management and phone texting technology to improve release's connections to care in the community.

This study will have extensive tracking of outcomes. The key outcome will be whether HIV infected participants receiving an intervention experience suppression of their viral load after release from jail . The investigators wish to demonstrate the ability to recruit participants into the SUCCESS intervention and repeatedly check community medical records to see how well their infection is being controlled after they linked to care. Investigators also want to conduct a survey at baseline, 3 months and 12 months.

Investigators will compare the viral load of participants receiving the intervention to participants passing through the jail who do not receive the outcome.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected (HIV+); age of or over 18 years;
* Mentally able to give consent; understand spoken English;
* Detained or sentenced in either the Fulton County Jail or the Atlanta City Detention Center; and
* Likely to leave within 6 weeks

Exclusion Criteria:

* Unable to give consent because of mental illness or inebriation;
* A recent participant in a randomized trial conducted by the investigators of an intervention to increase retention in HIV care (e.g., ARTAS)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2014-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
HIV viral load | 12 months after release from jail
  HIV viral load can be drawn; obtaining it shows that the person is in care. Ideally, it should be suppressed 12 months out of jail.
  One measurement of viral load within three months after release will demonstrate linkage; two clinical visits occurring within 12 months post release, with at least 2 clinical visits spaced a minimum of 3 months apart, will indicate retention.

SECONDARY OUTCOMES:
Show feasibility of conducting protocol | Four months
  Demonstrate that 14 persons can be recruited per month and that delivery of the intervention is feasible.

CONTACTS AND LOCATIONS:
Overall Officials: Anne C Spaulding, MD MPH, Principal Investigator — Emory University
Locations (1):
- Fulton County Jail, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Spaulding AC, Drobeniuc A, Frew PM, Lemon TL, Anderson EJ, Cerwonka C, Bowden C, Freshley J, Del Rio C. Jail, an unappreciated medical home: Assessing the feasibility of a strengths-based case management intervention to improve the care retention of HIV-infected persons once released from jail. PLoS One. 2018 Mar 30;13(3):e0191643. doi: 10.1371/journal.pone.0191643. eCollection 2018. PMID 29601591